CLINICAL TRIAL: NCT06123052
Title: A Descriptive Qualitative Study Using Semi-structured Individual Interviews to Get a Better Understanding of Patients' (un)Ability and (un)Willingness to Use IBD Care Everywhere (IBD-CE), a Telemonitoring Application for Patients With Inflammatory Bowel Diseases
Brief Title: A Qualitative Study on Patients' (un)Ability and (un)Willingness to Use Telemonitoring in Inflammatory Bowel Diseases
Status: Completed | Type: Observational
Sponsor: Franciscus Gasthuis (Other)
Collaborators: Jeroen Bosch Ziekenhuis (Other)
Responsible Party: Sponsor
Other Study IDs: 2023.07.06.01
Record Dates: First submitted 2023-08-08; First posted 2023-11-08 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Telemedicine; Inflammatory Bowel Diseases; Disparity; Health Equity
Keywords: UTAUT2; COM-B; Patient empowerment
MeSH Terms: conditions — Inflammatory Bowel Diseases; Patient Participation | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients not interested in IBD-CE: Interview
  Interventions: Other: Interview
- Patients interested in IBD-CE: Interview
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — This is a descriptive qualitative study using semi-structured individual interviews. The interview will aim to collect more information about the patients' underlying motives that influence their ability or willingness to use IBD-CE. An interview guide has been developed for this purpose, based on topics derived from the Unified Theory of Acceptance and Use of Technology (UTAUT) model, the COM-B model for behavioural change and the model of positive health. This interview guide is divided into four sections, each introduced by an initial question. Subsequent follow-up questions will be formulated based on the patients' responses.
  Furthermore, patient characteristics, disease characteristics, and socio-demographic data will be collected from the Electronic Medical Record (EMR). These data will provide insights into various aspects of the patients' profiles and are based on characteristics that seem to be determinants of technology acceptance and/or digital health literacy.

SUMMARY:
Crohn's disease and ulcerative colitis (inflammatory bowel disease, IBD) are chronic intestinal inflammations with considerable impact on quality of life. Due to the chronic nature of the disease and the complex treatment involving regular outpatient follow-up visits, IBD care places a substantial burden on both patients and the healthcare system. Providing appropriate care, as described in the National Integrated Care Agreement, is becoming increasingly important.

Telemonitoring is a promising alternative to conventional consultations, with evidence even suggesting improved quality of care. We have developed the telemonitoring application *IBD Thuis* to measure disease activity at home.

The aim of this study is to develop a more effective, safe, and patient-centered approach to telemonitoring, and to deliver the right care in the right place in line with the National Integrated Care Agreement. In this study, we investigate which patients are suitable for telemonitoring. Through interviews, we aim to gain insight into the factors that influence patients' willingness and ability to use telemonitoring, with specific attention to behavior change and technology acceptance.

DETAILED DESCRIPTION:
Introduction: Telemedicine has shown to play a promising role in improving IBD treatment. However, it remains uncertain which patients benefit from telemedicine. A feasibility and development project using IBD Care Everywhere (IBD-CE), a telemonitoring application, found that some patients were unable or unwilling to use the application. However, why patients were not able or willing to use the application remains unknown. The WHO global strategy aims to implement telemedicine while ensuring digital health equity. Concerns exist that telemedicine may exacerbate healthcare disparities.

Research question: The aim of this qualitative study is to get a better understanding of factors influencing patients' (un)ability and (un)willingness to use IBD-CE. These insights could help to offer the best individualised IBD care to patients. This led to the following research questions:

1. What influences patients' (un)ability or (un)willingness to use IBD Care Everywhere? 1.1 What are the distinguishing characteristics of patients (un)willing and (un)able to use IBD Care Everywhere? 1.2 How can we support patients in making an informed choice between telemonitoring and standard care?

Study design: This is a qualitative study using semi-structured interviews. Information about patient characteristics and potential factors that influence patients' ability or willingness to use IBD-CE will be collected. To guide the topics in the interview, three theories/models will be used:

1. The Unified Theory of Acceptance and Use of Technology (UTAUT) model
2. The COM-B model for behavioural change
3. The model of positive health Data will be analysed using thematic analysis.

Study population: Consecutive adult IBD patients (> 18 years) in stable remission, visiting the outpatient clinic at the Jeroen Bosch Hospital and Franciscus Gasthuis & Vlietland will be asked if they are willing to participate. Next, a total of 24 patients will be included through purposeful sampling. Both patients unwilling to use IBD-CE and patients interested in IBD-CE will be included. Should data saturation not have occurred, more patients will be included.

Expected results and relevance: Our objective is to get better insights in the motivations of patients to choose for telemonitoring or standard care. We aim to comprehend the requirements of patients to provide them with care that aligns with patients' needs.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years
* A confirmed IBD-diagnosis according to current guidelines
* Maintenance therapy with no medication changes in the last three months
* Remission:
* Crohn's disease: Faecal calprotectin (FCP) < 100 µ g/g and Harvey Bradshaw Index (HBI) < 5
* Ulcerative Colitis: Faecal calprotectin (FCP) < 250 µ g/g and Simple Clinical Colitis Activity Index scores (SCCAI) < 3

Exclusion Criteria:

* Presence of a stoma
* Presence of an ileo-anal pouch or ileorectal anastomosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise adult (>18 years) IBD patients visiting the outpatient clinics at Jeroen Bosch Hospital and Franciscus Gasthuis & Vlietland. These hospitals are teaching institutions with a combined patient population of approximately 4000 individuals.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Explorative data | through study completion, an average of 6 months
  Based on topics derived from the Unified Theory of Acceptance and Use of Technology (UTAUT) model, the COM-B model for behavioral change, and the model of positive health. This data is evaluated with the semi-structured interview

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Jeroen Bosch Ziekehuis, 's-Hertogenbosch
  - Franciscus, Rotterdam

IPD SHARING:
Plan to Share IPD: No